CLINICAL TRIAL: NCT01675505
Title: Psychological Well-being Outcomes in Disease-free Survivors of Colorectal Cancer Following Curative Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Antoniadis Diomidis, Phd student, Aristotle University Of Thessaloniki
Other Study IDs: Phd Antoniadis
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Adaptation, Psychological; Functional Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients: Inclusion criteria:
  Patients with first-diagnosed colon cancer. Age 18-60 y.o.
  Exclusion criteria:
  Metastatic colon cancer. Former psychiatric history. Substance use. Previous serious medical conditions.

SUMMARY:
The purpose of the study is to investigate whether there are prognostic factors regarding the mental and functional adjustment of colon cancer patients following curative surgery. Patients will be selected using specific inclusion criteria. Prognostic factors investigated include personality characteristics, initial distress, medical, social and economic factors. The utmost purpose of the study is to assist clinicians with the timely identification of vulnerable patients in order to ensure their proper management and their optimal adjustment.

Moreover this is the first study using the Distress Thermometer in Greek patients with cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with first-diagnosed colon cancer.
* Age 18-60 years

Exclusion Criteria:

* Metastatic colon cancer.
* Former psychiatric history.
* Substance use.
* Previous serious medical conditions.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Greek population from Northern Greece who are diagnosed with colon cancer for the first time and are admitted to the 1st Propedeutic Surgical Department of AHEPA General University Hospital of Thessaloniki for surgery.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2012-05

CONTACTS AND LOCATIONS:
Locations (1):
- Greece, 1st Propedeutic Surgical Department, AHEPA General University Hospital, Thessaloniki, Greece

REFERENCES:
- [Background] Jimmie C. Holland, William S. Breitbart, Paul B.Jacobsen, Marguerite S. Lederberg, Matthew J. Loscalzo, Ruth McCorkle. Psycho-oncology, second edition, Oxford University Press, 2010 National Comprehensive Cancer Network. Distress management. Clinical practice guidelines. J Natl Compr Canc Netw. 2003;1:344-74. Ward WL, Hahn EA, Mo F, Hernandez L, Tulsky DS, Cella D. Reliability and validity of the Functional Assessment of Cancer Therapy-Colorectal (FACT-C) quality of life instrument. Qual Life Res. 1999;8:181-95. Watson M, Law M, dos Santos M, Greer S, Baruch J, Bliss J. The Mini-MAC: further development of the Mental Adjustment to Cancer Scale. J Psychosoc Oncol1994;12:33-46.